CLINICAL TRIAL: NCT00204581
Title: Intralesional Treatment With Interleukin-2 (Proleukin) in Soft Tissue Melanoma Metastases. A Phase II, Prospective, Open, Multicenter Trial
Brief Title: Intralesional Treatment With Interleukin-2 (Proleukin) in Soft Tissue Melanoma Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Skin Cancer Programme, Dept. of Dermatology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL-2-LOK-MM
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2009-02

CONDITIONS: Melanoma
Keywords: Melanoma; Soft tissue metastases; Interleukin-2
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; aldesleukin

INTERVENTIONS:
Drug: Interleukin-2 (Proleukin) — 6-12 MIE/d 3times a week
  Other Names: Proleukin

SUMMARY:
The intra-/perilesional application of interleukin-2 seems to be a safe and effective treatment of skin and soft tissue metastases in malignant melanoma. Especially in case of intransit metastases the overall survival rate is still 20-30%.

However, the management of intransit metastases is sometimes difficult because of frequent recurrences. IL-2 intralesionally seems to be an non-invasive option as pilot studies indicate. In this study the safety and efficacy of IL-2 are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Informed consent
* Histologically proven melanoma
* Have confirmed stage IIIB or stage IV disease (AJCC 2002) with skin or soft-tissue metastases

Exclusion Criteria:

* Pregnant or lactating women
* Patients with severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina)
* Patients with severe liver disease or severe renal disease
* Simultaneous immunosuppressive treatment (e.g. steroids)
* Simultaneous chemotherapy
* Pretreated soft-tissue or skin metastases (e.g. cryo-, radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-08; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy in regard to complete and partial response | 4 weeks

SECONDARY OUTCOMES:
Overall survival | every 6 months
Side-effects | during treament and 4 weeks afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — Skin Cancer Program, Department of Dermatology, University Hospital Tübingen
Locations (1):
- Skin Cancer Program, Department of Dermatology, Liebermeisterstrasse 8, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Radny P, Caroli UM, Bauer J, Paul T, Schlegel C, Eigentler TK, Weide B, Schwarz M, Garbe C. Phase II trial of intralesional therapy with interleukin-2 in soft-tissue melanoma metastases. Br J Cancer. 2003 Nov 3;89(9):1620-6. doi: 10.1038/sj.bjc.6601320. PMID 14583759
- See also: Link to published abstract — http://www.ncbi.nlm.nih.gov/pubmed/20564107